CLINICAL TRIAL: NCT00791882
Title: Evaluation of Social Skills Training in Reducing Negative Symptoms in Patients With Refractory Schizophrenia
Brief Title: Social Skills Training in Refractory Schizophrenia
Acronym: SST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Helio Elkis MD PhD, Instituto de Psiquiatria da Faculdade de Medicina da Universidade de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SST
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Schizophrenia and Disorders With Psychotic Features
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group of behaviors by which someone express feelings, attitudes, wishes,opinions and rights , in an adequate manner regarding situation and context.
  Social skills are the substrate for social competence, which is the ability to find and legitimate relevant and personal goals
  Interventions: Behavioral: Social Skills Training
- 2 (No Intervention): Control group will attend the same number of sessions, but without intervention of the therapists
  Interventions: Behavioral: Social Skills Training

INTERVENTIONS:
Behavioral: Social Skills Training — A program developed during 20 weeks according to adapted BELLACK 's manual (1997),including sessions in group one hour per week.
  Other Names: Social Skills Training and Control group without active intervention.

SUMMARY:
Objective Primary:

To evaluate the efficacy of social skills training in reducing negative symptoms in patients with refractory schizophrenia, in comparison with control (befriending group).

Secondary:

To evaluate changes in social functioning.

To evaluate the effect of SST in other dimensions of psychopathology: positive symptoms, depression and general psychopathology.

To evaluate the impact of SST in cognition.

Hypothesis Social skills training is more effective than control group (Befriending) in reducing negative symptoms in patients with refractory schizophrenia.

DETAILED DESCRIPTION:
In schizophrenia positive symptoms can be improved with an antipsychotic treatment. However there is a subgroup of patients who have a predominance of persistent negative symptoms that do not respond to antipsychotic treatment, such as blunted affect , emotional and social withdrawal, and there is evidence that such symptoms can improve with psychosocial interventions.

The objective of this study is to evaluate the efficacy of Social Skills Training on negative symptoms in patients with refractory schizophrenia by means of a randomized, single-blind controlled trial with the duration of a year, including, follow up.

This study will be conducted in two groups: one group will receive social skills training (N=46) and a control group (N=46) will attend the same number of sessions, but without intervention of the therapists (befriending).

Psychiatric, psychological and neuropsychological aspects will be evaluated at baseline, after 20 weeks and 6 months after the end of the intervention.

The scales that will be used for the psychiatric assessments are: PANSS (reduction of 20% in the negative subscale), CGI, CALGARY, SDS, and PSP, As well as the Social Skills Inventory IHS. The neuropsychological assessment will have groups of scales to measure: Attention, Memory, Executive Functions, Estimated Intellectual Efficiency and a ToM. For statistical , the repeated measure ANOVA will be used, as well as the effect size and number needed to treat.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia can´t not be over 10 years old.
* Age between 18 and 55 years old.
* A minimum of 16 in negative subscale of PANSS.
* A score 4 in at least 3 of the following symptoms:

  * blunted affect
  * social withdrawal
  * rapport
  * passive social withdrawal
  * lack of spontaneity
  * motor retardation
  * active social avoidance
* Stable disease, in use of clozapine, without recent hospitalization.

Exclusion Criteria:

* Comorbid substance use.
* Axis I comorbidity.
* History of head trauma or neurological disease.
* Clinical problems which can affect central nervous system.
* Mental retardation.
* Patients treated with other antipsychotic than clozapine.
* Patients who underwent other psychosocial treatments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Response: at least 20% decrease at PANSS - negative subscale after 20 weeks, in comparison with baseline, maintained at 26 weeks follow-up. | 20 weeks treatment

SECONDARY OUTCOMES:
Improvement at PSP scores | 20 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Helio Elkis, MD PhD, Principal Investigator — Departamento de Psiquiatria da FMUSP
Locations (1):
- Instituto de Psiquiatria do HCFMUSP, São Paulo, São Paulo, Brazil